CLINICAL TRIAL: NCT07370285
Title: Enhancing Pediatric Nursing Students' Communication Skills and Grit Through an AI-Supported Empathy-Map Scaffolding Model: A Practice-Based Study
Brief Title: AI-Supported Empathy Mapping to Enhance Communication and Grit in Pediatric Nursing Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yu-Shiu Liu, Assistant Professor, Mackay Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25MMHIS511e
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Artificial Intelligence (AI); Empathy; Scaffolding; Pediatric Nursing; Communication Skills; Grit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 2（Control / Comparison Arm） (No Intervention)
- AI-Supported Empathy-Map Scaffolding Intervention (Experimental)
  Interventions: Behavioral: AI-Supported Empathy-Map Scaffolding Model

INTERVENTIONS:
Behavioral: AI-Supported Empathy-Map Scaffolding Model — The AI-Supported Empathy-Map Scaffolding Model is an educational intervention that combines empathy-map construction with AI-assisted reflective prompts to enhance communication skills, empathy, and grit in pediatric nursing students. The intervention uses case-based learning within regular coursework, involves no clinical treatment or patient contact, and is considered minimal risk.
  Arms: AI-Supported Empathy-Map Scaffolding Intervention

SUMMARY:
The nurse-patient communication environment in pediatric care is characterized by high uncertainty and complexity. Due to children's limited language development and emotional regulation abilities, coupled with parents' high level of involvement, nursing students often experience anxiety, lack of confidence, and avoidance behaviors, which negatively affect their clinical learning outcomes and the establishment of therapeutic relationships. Therefore, providing effective communication support strategies is essential in pediatric nursing education. This study aims to implement an instructional scaffolding model using artificial intelligence (AI)-generated empathy maps to enhance the communication skills, empathy performance, and grit of nursing students during pediatric clinical practicums when encountering communication challenges.

A mixed-methods research design was adopted, and the participants were third-year nursing students enrolled in a pediatric nursing practicum course. The teaching intervention included AI-assisted generation of age-appropriate communication strategies, the construction of a grit-oriented empathy map, small group scenario-based exercises, and the application of learned strategies in clinical settings. Quantitative data were collected using pre- and post-intervention assessments, including an empathy scale, a communication skills scale, and a grit scale, to evaluate changes in learning outcomes. Qualitative data, including reflective journals, clinical observations, and focus group interviews, were analyzed to explore students' learning processes and strategy adaptations. Triangulation was applied to strengthen the validity of the findings.

It is anticipated that this teaching model will enhance students' understanding of pediatric patients' emotional needs, strengthen their communication strategy application and clinical interaction quality, and promote persistence and adaptability in challenging situations. Through evidence-based teaching practice, this study is expected to provide a feasible and scalable innovative instructional model that supports the effective integration of AI into clinical nursing education, thereby improving pediatric nursing competence and the quality of care for children.

ELIGIBILITY:
Inclusion Criteria:

1. Undergraduate nursing students aged 18 years or older
2. Students enrolled in the Pediatric Nursing Practicum course

Exclusion Criteria:

1. Students who have not passed the Pediatric Nursing course

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-04-20 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Communication Skills | Baseline (pre-intervention) and immediately post-intervention
  Communication Competence Instrument (CCI). The Communication Competence Instrument was developed by Lee (2013) to enhance nurse-patient communication skills among nursing students. The instrument consists of eight items rated on a five-point Likert scale, with scores ranging from 1 (strongly disagree) to 5 (strongly agree). Sample items include: "I am able to establish a good nurse-patient relationship with patients/family members" and "I am able to ensure that patients/family members understand the key points of the communication." Higher scores indicate better communication competence.
  In Lee's study, the instrument demonstrated excellent reliability and validity, with a Cronbach's α of 0.92, a Spearman-Brown coefficient of 0.88, and a Guttman split-half coefficient of 0.88, indicating strong internal consistency and satisfactory psychometric properties for assessing communication behaviors.